CLINICAL TRIAL: NCT01067820
Title: Phase IIb Multi-center, Double-blind, Randomized, Parallel Group, Placebo-controlled Clinical Trial for the Assessment of Coronary Plaque Changes With RVX000222 as Determined by Intravascular Ultrasound
Brief Title: ApoA-I Synthesis Stimulation and Intravascular Ultrasound for Coronary Atheroma Regression Evaluation
Acronym: ASSURE I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Resverlogix Corp (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RVX222-CS-007
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Artery Disease
Keywords: ApolipoproteinA1; HDL-C; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — apabetalone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RVX000222, 200 mg daily (Experimental)
  Interventions: Drug: RVX000222
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo RVX000222

INTERVENTIONS:
Drug: RVX000222 — capsule, 200 mg, administer with food, 100 mg twice daily 10-12 hrs apart, 26 weeks
  Arms: RVX000222, 200 mg daily
Drug: Placebo RVX000222 — capsule, administer with food, twice daily 10-12 hrs apart, 26 weeks
  Arms: Placebo

SUMMARY:
This study is designed to characterize the early effects of ApoA-I synthesis with RVX000222 on coronary atherosclerotic disease when administered to patients with coronary artery disease and have a low HDL-C level, as assessed by Intravascular Ultrasound (IVUS) in addition to standard background therapy.

DETAILED DESCRIPTION:
One-third of the US population, almost 80 million adults, have cardiovascular disease and mortality associated with heart disease still remains as a leading cause of death around the world. The major risk factors for cardiovascular disease associated with atherosclerosis is dyslipidemia, characterized by high levels of low density lipoprotein (LDL) and/or low levels of high density lipoprotein (HDL). The widespread use of statins in patients at risk for cardiovascular disease has led to lower LDL levels but has had little effect on HDL levels. HDL has a well established role in atherosclerosis and cardiovascular disease protection. HDL mediates the removal of cholesterol from the atherosclerotic plaques for elimination from the body. The major component of HDL consists of apolipoprotein A-I (ApoA I). Recent intervention studies with synthetic HDL particles and recombinant ApoA-I have shown that HDL has the capacity to reverse coronary atherosclerosis. Increasing ApoA-I is likely to have a favorable effect on atherosclerotic plaque stability and size and on cardiovascular diseases. RVX000222 is a member of a novel class of small molecules that are candidates for the treatment of dyslipidemia by increasing plasma levels of HDL through increased ApoA-I transcription.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patient's >/= 18 years of age who are scheduled to undergo coronary angiography for a clinical indication.
2. Women of child-bearing potential, that is, women not surgically sterilized and between menarche and 1 year post menopause, must test negative for pregnancy at the time of enrollment based on a serum pregnancy test and agree to use a reliable method of birth control (for example, use of oral contraceptives or Norplant; a reliable barrier method of birth control (diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices; partner with vasectomy; or abstinence) during the study and for one month following the last dose of study drug.
3. Current (Local lab within 60 days prior to Visit 1). HDLC of </= 45 mg/dL (1.2 mmol/L) for females and HDLC of </=40 mg/dL (1.0 mmol/L) for males.
4. In the opinion of the investigator patients currently not on statin therapy will be able to start either atorvastatin (10 mg, 20mg or 40mg) or rosuvastatin (5mg, 10mg or 20 mg) at Visit 1.
5. In the opinion of the investigator patients currently on statin therapy other than atorvastatin (10 mg, 20mg or 40mg) or rosuvastatin (5mg, 10mg or 20 mg) can be switched to rosuvastatin (5mg, 10mg or 20 mg) at Visit 1.
6. Patients must meet all of the following criteria at the qualifying coronary catheterization procedure:

   A. Entire Coronary Circulation: Angiographic evidence of coronary heart disease as defined by at least one lesion in any of the three major native coronary arteries that has >20 percent reduction in lumen diameter by angiographic visual estimation or prior history of PCI. This vessel need not be the target coronary artery for IVUS. Any vessel with previous PCI may not be used as the target coronary artery.

   B. Left Main Coronary Artery: Must not have a >50 percent reduction in lumen diameter by visual angiographic estimation.

   C. Target Coronary Artery for IVUS: Must be accessible to the IVUS catheter. Must have a <50 percent reduction in lumen diameter by angiographic visual estimation throughout a segment of at least 40 mm in length (the "target segment"). A lesion of up to 60 percent stenosis is permitted, distal to the target segment. A single branch of the "target vessel" may have a narrowing up to but <70 percent by visual estimation, as long as the target segment contains no lesion >50 percent, provided that the branch in question is not a target for PCI or CABG. Has not undergone prior percutaneous coronary intervention or coronary artery bypass graft surgery. The target vessel is not currently a candidate for intervention or a likely candidate for intervention over the next 6 months. The target vessel may not be a bypass graft. The target vessel may not be a bypassed vessel. The target vessel may not be the culprit vessel for a previous MI.
7. Have given signed informed consent to participate in this study.

Exclusion Criteria:

1. Clinically significant heart disease which will require coronary bypass, PCI, cardiac transplantation, surgical repair and/or replacement during the course of the study.
2. Any elective surgical procedure that would require general anesthesia during the course of the study.
3. Coronary artery bypass graft (CABG) procedure within the past 90 days.
4. Previous or current diagnosis of severe heart failure (NYHA Class III-IV) or a documented left ventricular ejection fraction (LVEF) of <25 percent as determined by contrast left ventriculography, radionuclide ventriculography or echocardiography, the absence of an LVEF measurement in a patient without a previous or current diagnosis of heart failure does not prohibit entry into the study.
5. Patients with evidence of cardiac electrophysiologic instability including a history of uncontrolled ventricular arrhythmias, uncontrolled atrial fibrillation/flutter or uncontrolled supraventricular tachycardias with a ventricular response heart rate of >100 beats per minute at rest within 4 weeks prior to Visit 1.
6. Evidence of renal impairment as determined by any one of the following:

   * serum creatinine >1.5 mg/dL (>133 micromol/L) by central lab at Visit 1,
   * a calculated creatinine clearance less than 60 ml/min at Visit 1
   * a history of dialysis,
   * a history of nephrotic syndrome.
7. Have hypertension that is uncontrolled defined as 2 consecutive measurements of sitting blood pressure of systolic >160 mm Hg or diastolic >95 mm Hg at Visit 1.
8. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive beta-hCG laboratory test (>/= 5 mIU/mL).
9. Current or recent (within 12 month prior to Visit 1) treatment with immunosuppressants (eg, Cyclosporine).
10. Use of fibrates any dose or niacin/nicotinic acid 250 mg or more within 90 days prior to Visit 1.
11. Atorvastatin >40 mg daily at Visit 1.
12. Rosuvastatin >20 mg daily at Visit 1.
13. Triglycerides >400 mg/dL at Visit 1.
14. Any medical or surgical condition which might significantly alter the absorption, distribution, metabolism or excretion of medication including, but not limited to any of the following: cholecystitis, Crohn's disease, ulcerative colitis, or any gastric bypass alteration.
15. Evidence of hepatic disease as determined by any one of the following: a history of hepatic encephalopathy, history of Hepatitis B, C or E, history of esophageal varices, history of porta-caval shunt. Any one of the following liver enzymes that is >ULN by central lab at Visit 1: ALT, AST, GGT
16. A total bilirubin that is >ULN by central lab at Visit 1.
17. History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
18. History or evidence of drug or alcohol abuse within the last 12 months.
19. Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
20. Use of other investigational drugs and devices at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
21. History of noncompliance to medical regimens or unwillingness to comply with the study protocol.
22. Any condition that in the opinion of the investigator would confound the evaluation and interpretation of efficacy and/or safety data.
23. Persons directly involved in the execution of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The nominal change in percent atheroma volume (PAV) from baseline to 26 weeks postrandomization, as determined by intravascular ultrasound (IVUS) within the RVX000222 treated group. | baseline to 26 weeks postrandomization
  To evaluate the effect of RVX000222 on the change in burden of coronary atherosclerosis, as measured by percent atheroma volume (PAV), in patients with coronary artery disease and a low level of HDL-C requiring angiography for a clinical indication.

SECONDARY OUTCOMES:
Nominal change in percent atheroma volume (PAV), from baseline to 26 weeks postrandomization, as determined by intravascular ultrasound (IVUS) within the RVX000222 treated group compared to placebo. | baseline to 26 weeks postrandomization
  To evaluate the effect of RVX000222 on the change in total atheroma volume (TAV), changes in the 10-mm most diseased artery sub-segment containing the most amount of disease and the percentage of patients who demonstrate regression of coronary atherosclerosis.
Nominal change in total atheroma volume (TAV) from baseline to 26 weeks postrandomization, as determined by intravascular ultrasound (IVUS) in the RVX000222 treated group as well as compared to placebo. | baseline to 26 weeks postrandomization
  To evaluate the effect of RVX000222 on the change in total atheroma volume (TAV), changes in the 10-mm most diseased artery sub-segment containing the most amount of disease and the percentage of patients who demonstrate regression of coronary atherosclerosis.
Nominal change in total atheroma volume (TAV) for the 10-mm sub-segment with the greatest disease burden at baseline, within the RVX000222 treated group as well as compared to placebo. | baseline to 26 weeks postrandomization
  To evaluate the effect of RVX000222 on the change in total atheroma volume (TAV), changes in the 10-mm most diseased artery sub-segment containing the most amount of disease and the percentage of patients who demonstrate regression of coronary atherosclerosis.
Proportion of patients with regression of coronary atherosclerosis, defined as a change in percent atheroma volume (PAV) from baseline to 26 weeks of less than zero (i.e. any reduction in PAV). | baseline to 26 weeks postrandomization
  To evaluate the effect of RVX000222 on the change in total atheroma volume (TAV), changes in the 10-mm most diseased artery sub-segment containing the most amount of disease and the percentage of patients who demonstrate regression of coronary atherosclerosis.
Percent change from baseline in HDL-C, ApoA-I, and HDL-subclasses at various time points within the RVX000222 treated group as well as compared to placebo. | Week 14 and 26
  To evaluate the effect of RVX000222 on biomarkers (HDL-C, ApoA-I, HDL-subclasses) at various time points.
Incidence of adverse events by treatment group, including major adverse cardiac events (MACE) (death, MI, stroke, coronary revascularization, hospitalization for ACS or heart failure). | Continuous
  To evaluate the safety and tolerability of RVX000222.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nicholls, MBBS, PhD, Principal Investigator — Intravascular Ultrasound Core Lab, Cleveland Clinic
Locations (42):
- Argentina (5):
  - La Plata, Buenos Aires
  - Buenos Aires
  - Corrientes
  - Córdoba
  - San Isidro
- Belgium (4):
  - Brussels
  - Charleroi
  - Edegem
  - Genk
- Brazil (7):
  - Brasília
  - Cariacica
  - Curitiba
  - Goiânia
  - Porto Alegre
  - São Paulo
  - Uberlândia
- Hungary (3):
  - Budapest
  - Pécs
  - Szeged
- Netherlands (7):
  - Alkmaar
  - Amsterdam
  - Eindhoven
  - Enschede
  - Nijmegen
  - Rotterdam
  - Zwolle
- Poland (2):
  - Katowice
  - Warsaw
- Russia (4):
  - Moscow
  - Orenburg
  - Saint Petersburg
  - Tomsk
- Spain (10):
  - Badalona
  - Barcelona
  - Cartagena
  - Galdakao
  - Gijón
  - Madrid
  - Málaga
  - Santander
  - Santiago de Compostela
  - Vigo

REFERENCES:
- [Derived] Nicholls SJ, Puri R, Wolski K, Ballantyne CM, Barter PJ, Brewer HB, Kastelein JJ, Hu B, Uno K, Kataoka Y, Herrman JP, Merkely B, Borgman M, Nissen SE. Effect of the BET Protein Inhibitor, RVX-208, on Progression of Coronary Atherosclerosis: Results of the Phase 2b, Randomized, Double-Blind, Multicenter, ASSURE Trial. Am J Cardiovasc Drugs. 2016 Feb;16(1):55-65. doi: 10.1007/s40256-015-0146-z. PMID 26385396